CLINICAL TRIAL: NCT04064034
Title: Evaluation of the Diagnostic Potential a Lateral Flow Assay to Detect QSOX1 Peptide in Patients With or at Risk for Pancreatic Cancer
Brief Title: ALateral Flow Assay to Detect QSOX1 Peptide in Patients With or at Risk for Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Douglas O. Faigel, Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-004658
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Pancreas Cancer; Pancreas Cyst
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Subjects with pancreas cancer (Experimental): Subjects will have blood collected and tested for Quiescin Sulfhydryl Oxidase 1 (QSOX1) protein with the lateral flow assay (LFA).
  Interventions: Other: Lateral Flow Assay (LFA)
- Subjects with non-cancerous disorders (Experimental): Subjects will have blood collected and tested for Quiescin Sulfhydryl Oxidase 1 (QSOX1) protein with the lateral flow assay (LFA).
  Interventions: Other: Lateral Flow Assay (LFA)
- Subjects with pancreas cyst (Experimental): Subjects already undergoing biopsy of a pancreas cyst will have cyst fluid collected and tested for Quiescin Sulfhydryl Oxidase 1 (QSOX1) protein with the lateral flow assay (LFA).
  Interventions: Other: Lateral Flow Assay (LFA)

INTERVENTIONS:
Other: Lateral Flow Assay (LFA) — Test to detect the Quiescin Sulfhydryl Oxidase 1 (QSOX1) protein

SUMMARY:
Researchers have developed a new test to measure a protein QSOX1 that is found to be elevated in subjects with pancreas cancer. Researchers are looking to use this test to compare subjects with pancreas cancer and subjects without pancreas cancer to see if this test could be used to diagnosis pancreas cancer.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with biopsy-proven adenocarcinoma prior to receiving any therapy such as surgery, radiation or chemotherapy.
* Patients without pancreas cancer.
* Adult patients with benign pancreas disorders such as pancreatitis with imaging within 12 months (CT, MRI, EUS) documenting no cancer.
* Healthy adults with blood specimens in an existing biobank.
* Patients with pancreatic cystic lesions.
* Adult patients undergoing clinically indicated EUS-guided FNA biopsy of pancreatic cystic lesions.

Exclusion Criteria:

* Prior treatment for pancreas cancer.
* Unable or unwilling to give consent.

Min Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Quiescin Sulfhydryl Oxidase 1 (QSOX1) in the blood | Baseline
  Number of subjects with the presence and concentration of QSOX1 peptide found in the blood samples by the lateral flow assay (LFA) test

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Faigel, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials